CLINICAL TRIAL: NCT05988242
Title: Effect of Primrose Oil Versus Lavender Oil on Hot Flashes and Night Sweats Among Menopausal Women
Brief Title: Effect of Lavender Versus Primrose Oil on Menopause Symptom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Zaghloul, Lecturer of maternal and newborn health nursing, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Lavender and Primrose
Record Dates: First submitted 2023-07-20; First posted 2023-08-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Menopause Syndrome
Keywords: Hot Flashes; Sweat; Menopause; Lavandula; Primula
MeSH Terms: conditions — Hot Flashes | interventions — evening primrose oil; lavender oil

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial will be used to fulfill the aim of proposed study. The randomized control trial (RCT) is a trial in which subjects are randomly assigned to one of two or more groups: the intervention (group A) who will receive evening primrose oil, the intervention (group B) who will receive lavender oil, the third group ( C) who will receive placebo (Spieth et al, 2016).
Who Masked: Participant, Investigator
Masking Description: Regarding the nature of the intervention it will be double blind as the women will not know which intervention will take and the randomization of the groups will be done by person other than the researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- primrose oil (Experimental): primrose oil
  Interventions: Other: Primrose oil
- lavender oil (Experimental): lavender oil
  Interventions: Other: Lavender oil
- the placebo group (Placebo Comparator): took the same bottle of oil which didn't contain the active substances but have the same shape, same oder, same color.
  Interventions: Other: placcebo

INTERVENTIONS:
Other: Primrose oil — group A will take primrose oil
  Arms: primrose oil
Other: Lavender oil — group B will take lavender oil
  Arms: lavender oil
Other: placcebo — this is the comparator group who will take the same bottle of oil which dosnt contain the active substances but have the sampe shape, same oder, same color
  Arms: the placebo group

SUMMARY:
there is a scanty of researches which integrate to investigate the comparing effect of evening primrose oil and lavender as the essential oil that affects on menopausal vasomotor symptoms especially hot flashes and night sweet Therefore, the current study is expected to contribute to the knowledge and practice regarding the effect of lavender versus primrose oil on hot flashes and night sweat in menopausal women.

DETAILED DESCRIPTION:
The aim of this study is to assess the efficacy of primrose oil versus lavender oil on hot flashes and night sweats among menopausal women

Research Hypotheses To fulfill the aim of this study the following research hypotheses will be formulated H1: Menopausal women who will receive evening primrose oil may show decrease in frequency and severity of hot flashes and night sweat as compared to those who will receive routine care H2: Menopausal women who will receive lavender oil may show decrease in frequency and severity of hot flashes and night sweat as compared to those who will receive routine care H3: There is a difference between menopausal women who will receive evening primrose oil versus lavender oil in relation to frequency and severity of hot flashes and night sweat Outcome measures

Sample A total of (150) menopausal women who will attend the out patient gynaecological clinic at Obstetrics and Gynecological hospital in Cairo university hospitals, Kasr El Ainy will be recruited for this study and randomly assigned to either group who will receive primrose oil (50) women, the other group who will receive lavender oil (50) women, the placebo group (50) who will take package of oil but dosnt contain the active substance .

Tools for Data Collection To fulfill the aim of the study fourth tools will be utilized for data collection. The first one the interviewing questionnaire which was designed by the researcher through extensive review of literature; the second tool is Daily hot flash / night sweets diaries; the third tool is Hot-flush/ night sweet problem-rating (HFNS Problem Rating) and the fourth tool is Hot Flash Related Daily Interference Scale (HFRDIS).

Tools used in the Randomized Control Trail:

First tool: Interviewing Questionnaires Schedule (Appendix A) This tool designed by the researcher after extensive literature review which constituted of four parts; first part data related to demographic characteristics such as age, level of education, residence and occupation. Second part data related to menstrual history and menopausal status.

Second tool: Daily hot flash / night sweets diaries Daily Hot Flash Diary: It is a selfreport dairy , in which participants recorded how many hot flashes they experienced on a daily basis as well as the severity of each hot flash on a scale of 1-3 (1 being mild, 2 moderate, and 3 severe). Hot flashes throughout a 7-day period were added to produce a weekly hot flash frequency score. While the number of hot flashes reported in each severity level was used to calculate the daily severity score, the total number of daily severity scores over the course of seven days was used to determine the hot flash severity index The hot flash severity score for each day was calculated as the sum of the number of hot flashes within each severity category, multiplied by the severity score for that category, with the resulting sum divided by the total number of hot flashes Third tool: Hot-flush/ night sweet problem-rating (HFNS Problem Rating) This tool is standardized tool to measure the extent to which HFNS are a problem, it is a subscale of the Hot Flush Rating Scale (HFRS) this validated self-report measure has three questions using 10-point Likert scales to rate the extent to which HFNS are problematic, distressing, and the cause of interference in daily life. Problem rating is calculated as the mean of the three questions, with higher scores indicating more problematic. This tool has significant correlations with diary recordings for hot flushes (r=0.97, p<0.001) and night sweats (r=0.94, p<0.001). HFRS has good test-retest reliability (r=0.8) and internal consistency (alpha=0.87); the internal reliability alpha coefficients 0.84. it is significantly associated (r=0.61-0.85 p<0.001) .

Fourth tool: Hot Flash Related Daily Interference Scale (HFRDIS) It is a 10-item scale to assess the degree to which hot flashes interfere with women's daily life activities. The first nine items assess the quality of daily life activities including work, social activities, leisure activities, sleep, mood, concentration, relationships with others, sexuality, and enjoyment of life and the tenth item assesses the overall quality of life. On a scale of 0 (do not interfere) to 10 (totally interfere), Women rate the extent to which hot flashes interfered with each item throughout the previous week. A total score is calculated by summing items. Higher scores reflect more interference from hot flashes and a greater impact on quality of life. The total score ranges from 0-100. This score was interpreted to the Mild interference 0-33•corresponding daily interference as follows: Moderate interference 34-67• Severe interference 68-100• Validity and reliability

Tools of data collection are standardized tool..UN standardized tools were submitted to 3 experts in the field of maternity nursing to test content validity, clarity of sentences and an appropriateness of content. Modifications were carried out according to the expert judgment before seeking the acceptance of ethical committee.

Ethical consideration An official approval to conduct the proposed study will be obtained from the Research Ethics Committee at faculty of nursing - Cairo University. As well, an official permission will be taken from the administrative personnel in the recommended settings. Also, each woman will be informed orally about the purpose of the trial and its importance. In addition, informed written consent will be obtained from women who will be willing to participate in the trial after ensuring that their participation in the trial will be voluntary and can be withdrawing at any time. As well as the anonymity, confidentiality and privacy of the information will be maintained.

ELIGIBILITY:
Inclusion Criteria:

* can read and write
* experienced amenorrhea for > 6 months
* mild or moderate-to-severe hot flashes at least twice daily
* normal blood pressure
* normal kidney and liver function
* no abnormal vaginal bleeding
* no sensitivity to herbal substances

Exclusion Criteria:

* Women with serious disease such as kidney, liver, seizure and allerg
* use of hormonal medications or herbal treatment in the preceding 2 months for treatment of hot flushes or night sweet

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
frequency of hot flashes among menopausal women. | Before intervention, 4 week after intervention, 8 week after intervention
  it will be assessed by Daily Hot Flash Diary: It is a selfreport dairy in which participants recorded how many hot flashes they experienced on a daily basis. Hot flashes throughout a 7-day period were added to produce a weekly hot flash frequency score
severity of hot flashes among menopausal women | Before intervention, 4 week after intervention, 8 week after intervention
  it will be assessed by Daily Hot Flash Diaryas well as the severity of each hot flash on a scale of 1-3 (1 being mild, 2 moderate, and 3 severe). the number of hot flashes reported in each severity level was used to calculate the daily severity score, the total number of daily severity scores over the course of seven days was used to determine the hot flash severity index.
  The hot flash severity score for each day was calculated as the sum of the number of hot flashes within each severity category, multiplied by the severity score for that category, with the resulting sum divided by the total number of hot flashes
to To what extent hot flash and night sweet are a problem | Before intervention, 4 week after intervention, 8 week after intervention
  This tool is standardized tool to measure the extent to which hot flash and night sweet are a problem, it is a subscale of the Hot Flush Rating Scale (HFRS) this validated self-report measure has three questions using 10-point Likert scales to rate the extent to which HFNS are problematic, distressing, and the cause of interference in daily life. Problem rating is calculated as the mean of the three questions, with higher scores indicating more problematic

SECONDARY OUTCOMES:
Hot Flash Related Daily Interference | Before intervention, 4 week after intervention, 8 week after intervention
  It is a 10-item scale developed by Carpenter, (2001) to assess the degree to which hot flashes interfere with women's daily life activities. The first nine items assess the quality of daily life activities including work, social activities, leisure activities, sleep, mood, concentration, relationships with others, sexuality, and enjoyment of life and the tenth item assesses the overall quality of life. On a scale of 0 (do not interfere) to 10 (totally interfere), Women rate the extent to which hot flashes interfered with each item throughout the previous week. A total score is calculated by summing items. Higher scores reflect more interference from hot flashes and a greater impact on quality of life. The total score ranges from 0-100. This score was interpreted to the Mild interference 0-33•corresponding daily interference as follows: Moderate interference 34-67• Severe interference 68-100•

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa Saad, lecturer, Study Chair — faculty of nursing
Locations (1):
- Faculty of nursinf, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the data will be shared online
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: four month
Access Criteria: will be published on magazine

REFERENCES:
- [Background] Kazemi F, Masoumi SZ, Shayan A, Oshvandi K. The Effect of Evening Primrose Oil Capsule on Hot Flashes and Night Sweats in Postmenopausal Women: A Single-Blind Randomized Controlled Trial. J Menopausal Med. 2021 Apr;27(1):8-14. doi: 10.6118/jmm.20033. PMID 33942584
- [Background] Farzaneh F, Fatehi S, Sohrabi MR, Alizadeh K. The effect of oral evening primrose oil on menopausal hot flashes: a randomized clinical trial. Arch Gynecol Obstet. 2013 Nov;288(5):1075-9. doi: 10.1007/s00404-013-2852-6. Epub 2013 Apr 27. PMID 23625331
- [Background] Reddi KK. Human granulocyte ribonuclease. Biochem Biophys Res Commun. 1976 Feb 23;68(4):1119-25. doi: 10.1016/0006-291x(76)90312-0. No abstract available. PMID 5077
- [Background] Baker FC, Lampio L, Saaresranta T, Polo-Kantola P. Sleep and Sleep Disorders in the Menopausal Transition. Sleep Med Clin. 2018 Sep;13(3):443-456. doi: 10.1016/j.jsmc.2018.04.011. PMID 30098758
- [Background] Carreiras M, Seghier ML, Baquero S, Estevez A, Lozano A, Devlin JT, Price CJ. An anatomical signature for literacy. Nature. 2009 Oct 15;461(7266):983-6. doi: 10.1038/nature08461. PMID 19829380
- [Background] Mehrpooya M, Rabiee S, Larki-Harchegani A, Fallahian AM, Moradi A, Ataei S, Javad MT. A comparative study on the effect of "black cohosh" and "evening primrose oil" on menopausal hot flashes. J Educ Health Promot. 2018 Mar 1;7:36. doi: 10.4103/jehp.jehp_81_17. eCollection 2018. PMID 29619387
- [Background] Green MR, Pastewka JV. The cationic carbocyanine dyes Stains-all DBTC, and Ethyl-Stains-all, DBTC-3,3',9 triethyl. J Histochem Cytochem. 1979 Mar;27(3):797-9. doi: 10.1177/27.3.90067.
- [Result] Tsai J, Chung YC, Chen FP, Yeh ML. [Effect of Aromatherapy on Menopausal Symptoms, Heart Rate Variability, and Sleep Quality in Women]. Hu Li Za Zhi. 2020 Feb;67(1):44-54. doi: 10.6224/JN.202002_67(1).07. Chinese. PMID 31960396
- [Result] Kazemzadeh R, Nikjou R, Rostamnegad M, Norouzi H. Effect of lavender aromatherapy on menopause hot flushing: A crossover randomized clinical trial. J Chin Med Assoc. 2016 Sep;79(9):489-92. doi: 10.1016/j.jcma.2016.01.020. Epub 2016 Jul 4. PMID 27388435